CLINICAL TRIAL: NCT05955144
Title: Clinical Validation of the Screening Tool Picterus Jaundice Pro to Assess Neonatal Jaundice Using Different Types of Smartphones
Brief Title: Clinical Validation of the Screening Tool Picterus JP Using Different Smartphones
Acronym: allphones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Picterus AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: allphone
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Repeatable bilirubin measurement independent of phone (Other): all subjects will receive bilirubin measurement from 4 different smartphones and a transcutaneous device to ensure that the measurement of bilirubin is not affected by phone camera
  Interventions: Device: Picterus JP

INTERVENTIONS:
Device: Picterus JP — Use Picterus Jaundice Pro, a smartphone app that is used to take photo of the newborns skin, where the Picterus calibration card is placed.

SUMMARY:
The overall aim of this study is to verify the quality of our internal developed camera validation systems and allow the use of Picterus JP on all smartphones.

DETAILED DESCRIPTION:
The overall aim of this study is to verify the quality of our internal developed camera validation systems and allow the use of Picterus JP on all smartphones.

Picterus JP bilirubin estimates from a Samsung S7 will be compared with three smartphones with different camera types and a TcB measurement The clinical outcomes will be compared to our camera validation systems. Skin color measurements using a spectrophotometer will be used for technical optimization of the camera validation system

ELIGIBILITY:
Inclusion Criteria:

* Infants born with gestational age > 37 weeks.
* Birth weight ≥ 2500 grams
* Age 1 - 14 days

Exclusion Criteria:

* Infants showing signs of inborn disease.
* Infants with skin rash or other skin disease that affects the skin where measurements are performed.
* Infants transferred to the pediatric ward for medical treatment.
* Infants that have received phototherapy in the last 24 hours

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
jaundice screening | 6 months
  reproducible jaundice screening independent of smartphone used

CONTACTS AND LOCATIONS:
Locations (1):
- St Olav Hospital, Trondheim, Norway